CLINICAL TRIAL: NCT02955420
Title: A Three-part, Randomized Study to Investigate the Safety, Tolerability, Pharmacokinetics and Efficacy of BC 007 in Healthy, Young Subjects and Elderly Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Efficacy of BC 007 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Berlin Cures GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBC007C101; 2015-005236-18 (EudraCT Number)
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
Keywords: Autoantibodies; Heart Failure; Fatigue Syndrome, Chronic; Idiopathic Pulmonary Hypertension; Cardiomyopathies
MeSH Terms: conditions — Heart Failure; Fatigue Syndrome, Chronic; Familial Primary Pulmonary Hypertension; Cardiomyopathies | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- BC 007 (15, 50, 150, 300, 450, 750, 1350, 1200 mg) (Experimental): Part A:
  BC 007 at doses of 15, 50 and 150 mg or matching placebo administered as i.v. bolus + infusion of 20 min (Cohorts 1 to 4). The sentinel pair of each cohort will be dosed without bolus.
  NaCl 0.9% (matching placebo) administered as i.v. bolus + infusion of 20 min (Part A: Cohorts 1 to 4).
  Part B:
  BC 007 at doses of 50 and 150 mg administered (Cohort 1) or a single dose < 50 mg or 150 mg (Cohort 2) as i.v. bolus + infusion of 20 min is administered to GPCR autoantibody positive subjects. The first subject in each dosing period of Cohort 1 will be dosed without bolus.
  Part C:
  BC007 administered at doses of 300 mg (Cohort 1), 450 mg (Cohort 2), 750 mg (Cohort 3), 1350 mg (Cohort 4) as i.v. bolus + infusion of 40 min to GPCR autoantibody positive subjects. The first three subjects in each dosing period of Cohort 1-4 will be dosed without bolus. In Cohort 5 BC007 dose of 1200 mg will be administered as a continuous infusion of 20 min.
  Interventions: Drug: BC 007; Drug: NaCl 0.9 %

INTERVENTIONS:
Drug: BC 007
Drug: NaCl 0.9 %

SUMMARY:
Berlin Cures develops BC 007 to treat patients suffering from diseases (chronic heart failure, pulmonary hypertension, chronic fatigue syndrome etc.) which are associated with functional autoantibodies (AAB) directed against G-protein coupled receptors (GPCR).

The first part of the study (part A) is designed to evaluate the safety and tolerability of ascending doses of BC 007. The study part is blinded and placebo controlled in order to better discriminate possible safety signals. The assessment of safety and tolerability in an elderly cohort is a bridge to dosing elderly GPCR AAB positive subjects in part B. The subjects in part A are confirmed to be GPCR AAB negative.

The objective of the second part of the study (part B) is to evaluate the efficacy of BC 007 in neutralizing AAB against GPCR shortly after dosing compared to baseline and to find the optimal dose for the neutralization of the AAB in all individuals. This dose shall be taken to progress into a Phase II/III trial with beta1-adrenergic receptor-AAB positive patients suffering from chronic heart failure.

DETAILED DESCRIPTION:
Part A

Primary objective is:

* To assess safety and tolerability of BC 007 after a single ascending intravenous (i.v.) bolus + infusion in healthy, young and elderly subjects.

Secondary objectives are:

* To determine the pharmacokinetic plasma and urine profiles of BC 007 in healthy, young and elderly subjects.

Part B

Primary objective is:

* To assess the neutralizing potency of BC 007 against GPCR autoantibodies alpha -1 adrenergic receptor, beta-1 adrenergic receptor, beta-2 adrenergic receptor or endothelin-A-receptor following ascending i.v. bolus + infusion.

Secondary objectives are:

* To assess safety and tolerability of BC 007 after a single ascending i.v. bolus + infusion in GPCR AAB (α(1)-adrenergic receptor AAB, ß(1)-adrenergic receptor AAB, ß(2)-adrenergic receptor AAB or endothelin-A-receptor AAB) positive healthy elderly subjects.
* To determine the pharmacokinetic plasma and urine profiles of BC 007 in GPCR AAB (α(1)-adrenergic receptor AAB, ß(1)-adrenergic receptor AAB, ß(2)-adrenergic receptor AAB or endothelin-A-receptor AAB) positive healthy elderly subjects.

Part C

Primary Objective

* To assess the neutralizing potency of BC 007 against GPCR autoantibodies alpha-1 adrenergic receptor (α(1)-AR AAB), beta-1 adrenergic receptor (ß(1)-AR AAB), beta-2 adrenergic receptor (ß(2)-AR AAB) or endothelin-A-receptor (ETA AAB) following ascending i.v. bolus + infusion.

Secondary Objectives

* To assess safety and tolerability of BC 007 after a single ascending i.v. bolus + infusion in GPCR AAB (α(1)-AR AAB, ß(1)-AR AAB, ß(2)-AR AAB or ETA AAB) positive healthy elderly subjects.
* To determine the pharmacokinetic plasma and urine profiles of BC 007 in GPCR AAB (α(1)-AR AAB, ß(1)-AR AAB, ß(2)-AR AAB or ETA AAB) positive healthy elderly subjects.

Explorative Objective

* To investigate the pharmacokinetic plasma and urine profiles of BC 007 metabolites in GPCR AAB (α(1)-AR AAB, ß(1)-AR AAB, ß(2)-AR AAB or ETA AAB) positive healthy elderly subjects

ELIGIBILITY:
Inclusion Criteria (main):

1. The subject is a healthy, male, non-smoker or slight/occasional smoker (less than or equal to 10 cigarettes per day), 18 to 45 years of age (Cohorts 1 to 3, Part A).
2. The subject is a healthy, male or female, non-smoker or slight/occasional smoker (less than or equal to10 cigarettes per day), 55 to 70 years of age (Cohort 4 [only in Part A] and Part B).
3. Female subjects are postmenopausal (verified by an appropriate serum FSH level and amenorrhea for at least one year).
4. The subject has a body mass index (BMI) range of 18.5 to 29.9 kg/m2 inclusive, (healthy young males as well as elderly subjects) and weighs at least 50 kg and < 100 kg.
5. The subject is positive for either one or the combination of GPCR α(1)- adrenergic receptor AAB, ß(1)-adrenergic receptor AAB, ß(2)-adrenergic receptor AAB and endothelin-A-receptor AAB (Part B only) at (pre-) screening prior to enrolment.
6. The subject is negative for GPCR α(1)-adrenergic receptor AAB, ß(1)-adrenergic receptor AAB, ß(2)-adrenergic receptor AAB and endothelin-A-receptor AAB at (pre-)screening prior to enrolment (Part A only).
7. Coagulation variables, uric acid, ALT, AST, alkaline phosphatase (ALP), GGT, bilirubin and creatinine must be within the normal laboratory reference ranges at screening.
8. Thyroid-stimulating hormone (TSH) must be within the normal laboratory reference range at screening.

Exclusion Criteria (main):

1. Any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic (specifically gout), urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, as judged by the Investigator.
2. Any history or current intake of beta blockers.
3. Any history of allergic reactions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 24 hours post dose
Part B: Conversion rate from positive GPCR AAB to negative immune status | 24 hours post dose
Part C: Conversion rate from positive GPCR AAB to negative immune status | 24 hours and 8-12 days post dose

SECONDARY OUTCOMES:
Part A, B and C: Area under the plasma concentration time curve (AUC) from time zero to the last quantifiable concentration (AUC0-t) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: Area under the plasma concentration time curve (AUC) from time zero extrapolated to infinity (AUC0-inf) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: AUC from time zero to 24 hour post-dose (AUC0-24) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: Maximum observed plasma concentration (Cmax) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: Apparent terminal half-life (t1/2) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: Nominal time of Cmax (tmax) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: Plasma clearance (CL) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: Volume of distribution during terminal phase (Vz) derived from BC 007 plasma concentrations | 24 hours post dose
Part A, B and C: Terminal elimination rate constant (λz) derived from BC 007 plasma concentrations | 24 hours post dose
A, B and C: Cumulative amount of unchanged drug excreted into urine (Ae) | 24 hours post dose
A, B and C: Fraction of intravenous administered drug that is excreted unchanged in urine (fe) | 24 hours post dose
Part A, B and C: Renal clearance (CLR) of BC 007 | 24 hours post dose
Part A, B and C: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Angela Sinn, Dr., Principal Investigator — Parexel
Locations (1):
- PAREXEL International GmbH, Early Phase Clinical Unit Berlin, Berlin, Germany

REFERENCES:
- [Derived] Becker NP, Haberland A, Wenzel K, Gottel P, Wallukat G, Davideit H, Schulze-Rothe S, Honicke AS, Schimke I, Bartel S, Grossmann M, Sinn A, Iavarone L, Boergermann JH, Prilliman K, Golor G, Muller J, Becker S. A Three-Part, Randomised Study to Investigate the Safety, Tolerability, Pharmacokinetics and Mode of Action of BC 007, Neutraliser of Pathogenic Autoantibodies Against G-Protein Coupled Receptors in Healthy, Young and Elderly Subjects. Clin Drug Investig. 2020 May;40(5):433-447. doi: 10.1007/s40261-020-00903-9. PMID 32222912